CLINICAL TRIAL: NCT06680401
Title: The Evaluation of Cytokines and Hormones as Biomarkers for Epithelioid Haemangioendothelioma and Generation of Patient-derived Preclinical Models to Assess the Activity of Anticancer Agents and Validate Novel Therapeutic Targets
Brief Title: Epithelioid Haemangioendothelioma Observational Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: EHE
Record Dates: First submitted 2024-03-20; First posted 2024-11-08 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-07

CONDITIONS: Clinical Presentation; Natural History; Treatment Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A: Patients newly diagnosed with advanced EE starting active surveillance
- Group B: Patients with new diagnosis of advanced, evolving EE, worthy of medical treatment
- Group C: Patients with a previous diagnosis of advanced EE, already under active surveillance
- Group D: Patients with a previous diagnosis of advanced EE with ongoing medical treatment
- Group E: Patients with localized EHE

SUMMARY:
The EHE observational study was developed to obtain a high number of datas such as clinical presentation, natural history, and treatment outcomes, cto identificate cytokines and hormones as biomarkers and generate patient-derived preclinical models as a tool to assess the activity of anticancer agents and validate novel therapeutic targets

DETAILED DESCRIPTION:
Epithelioid hemangioendothelioma (EHE) is an ultra-rare (incidence rate < 1/1000.000), translocated, vascular soft tissue sarcoma. It shows a pick of incidence in the 4th decade of life, and it is more commonly diagnosed in females, with reported disease onset during pregnancy.

Two specific translocations have been identified in EHE, representing an hallmark in diagnosis today: the fusion of Transcriptional Co-activator with a PDZ-motif (TAZ) with Calmodulin Binding Transcription Activator 1 (CAMTA1) which is present in almost 90 % of cases, and the fusion of Yes-associated Protein (YAP) and Transcription Factor E3 (TFE3) genes (YAP-TFE3), which can be found in around 10% of the patients. YAP and TAZ are well-defined downstream effectors in the Hippo pathway. Forced activation of YAP/TAZ is thought to drive EHE and contribute to key aspects of the cancer phenotype, including metastasis and fibrosis.

Most of the times, EHE presents as multifocal or metastatic at diagnosis, with lung, liver and bone being the more commonly involved. The clinical course ranges from cases naturally stable over time to those highly aggressive and rapidly fatal. Pleural effusion, lymph node metastases and pathologic features (nuclear pleomorphism, mitotic figures and presence of necrosis) have been reported to be associated with a worse outcome, but biological and molecular predictors are still lacking. In particular, there is a subgroup of EHE presenting with serosal involvement, typically associated with chronic mild fever, weight loss, asthenia, anorexia, severe disease- related pain, (more responsive to anti-inflammatory pain killers that morphine), and dyspnoea which seems to perform very poorly. The biological basis sustaining this presentation is completely unknown.

As of today, there are no reports available in literature providing a comprehensive description of the peculiar EHE radiological features, both for primary and metastatic disease at different sites, and their potential prognostic role has not been explored. In addition, there are no published data to indicate the optimal routine follow-up policy of surgically treated EHE patients with localised disease and the routine follow-up schedules differ across institutions. The appropriate frequency of imaging in cases suffering of distant metastases is also left to be determined.

Also, the definition of radiological progression and the assessment of treatment response in EHE remain major challenges. The appearance or worsening of serosal effusion, the changes in serosal involvement and the limited increase in size over a short-time interval in slow-growing variants are not promptly captured by Response Evaluation Criteria for Solid Tumor (RECIST) definition for disease progression. This makes the use of such criteria unsatisfactory in this complex disease and could potentially lead to a delay in progression recognition and treatment start. Similarly, being frequently observed in EHE under treatment, improvement of serosal effusion, reduction in size <30%, and correlation between radiology and symptoms should be taken into account when assessing treatment response.

Surgery is the mainstay of care in the local setting. Active surveillance can be a reasonable strategy for patients with naturally stable or asymptomatic, slowly progressive disease, reserving medical treatment to symptomatic or progressive cases.

Data on conventional chemotherapy in advanced EHE are limited to case reports and single-institution experiences and suggest a limited role for the drugs commonly used in adult-type soft tissue sarcomas. Signs of activity have been reported with the use of anti-angiogenics, including pazopanib, sorafenib, bevacizumab, alone or in combination with chemotherapy, and apatinib. Due to the peculiar natural history of the disease, the value of antiangiogenics and/or immunomodulatory agents has also been explored, with responses described with sirolimus, thalidomide, interferon, and celecoxib.

In absence of any active treatment available, EHE is a neglected disease, and the identification of new potentially active compounds, especially for patients affected by the more aggressive EHE variant. To this end, it looks to be of major importance to identify what is behind disease progression, the "inflammatory-like" disease presentation, and the prevalence of the disease in the female young population.

Several lines of evidence have highlighted the significance of inflammation at the local and/or systemic level in human tumor pathobiology. Indeed, inflammation can influence tumor progression, metastasis and therapeutic outcome by establishing a tumor supportive immune microenvironment. These processes are mediated through a variety of cytokines and hormones that exert their biological actions either locally or distantly via systemic circulation.

Estrogen signaling is mediated via several receptor proteins. In addition to the classical ERα and ERβ, the membrane-bound G-protein coupled estrogen receptor (GPER) mediates both the genomic and non-genomic effects of estrogen and has been implicated in the development of other tumors such as breast cancer. Interestingly, GPER stimulation activates YAP and TAZ as key effectors of the Hippo pathway. Insulin-like growth factor-1(IGF-1) has also been shown to regulate GPER expression and function, suggesting a crosstalk between growth factors and ERs The availability of translatable preclinical models of human EHE, able to properly recapitulate tumor biology and response to treatment of the clinical tumors, appears instrumental for the development of innovative and effective treatments. Patient-derived xenograft (PDX) models preserve the original histomorphological and molecular characteristics of the originating clinical tumors. We previously demonstrated the consistency between preclinical data obtained on PDXs of different soft-tissue sarcoma histotypes (solitary fibrous tumor, epithelioid sarcoma and dedifferentiated liposarcoma) and clinical results concerning the activity of several cytotoxic and molecularly targeted drugs, providing novel insight into the antitumor effect of different combinations that was instrumental to design novel clinical trials.

MicroRNAs (miRNAs) are small non-coding RNAs that negatively regulate gene expression at the post-transcriptional level. Their proven deregulation in several types of human cancer, and the possibility to be reliably detected in both tissue and blood specimens, have prompted the assessment of miRNAs as novel cancer biomarkers21. No information is currently available on miRNA expression and function in EHE.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of EHE according to 2020 WHO classification, performed on biopsy or surgical specimen
* Signed informed consent
* Adequate patient compliance to treatment or follow up
* No age limit

Exclusion Criteria:

* Impossibility to ensure adequate compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to include at least 50 patients (range: 50-70) in 36 months, followed by a follow up time of 3 years.68 including The Royal Marsden Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Demographic description | Through study completion, an average of 1 year
  To provide a demographic description of the population affected by advanced EHE
Patient status | Through study completion, an average of 1 year
  To provide a description of clinical presentation, natural history, and treatment pattern in patients with advanced EHE
Tumor-related symptoms | Through study completion, an average of 1 year
  To provide a description of tumour-related symptoms and their changes over time
Tumor-related pain | Through study completion, an average of 1 year
  To provide a tumor-related pain assessment
Clinical prognosis | Through study completion, an average of 1 year
  To prospectively identify clinical prognostic and predictive factors
radiological features | Through study completion, an average of 1 year
  To describe the radiological features of the disease (group A, B, C, D, E)
correlation between radiological features and outcome | Through study completion, an average of 1 year
  To correlate radiologic features with the outcome and the tested plasma levels of the cytokines and hormones (group A, B, C, D, E)
radiological response and systemic treatment | Through study completion, an average of 1 year
  To assess radiologic response to systemic treatments by basing on RECIST 1.1 assessment (group B, D).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stacchiotti, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS IstitutoNazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sardaro A, Bardoscia L, Petruzzelli MF, Portaluri M. Epithelioid hemangioendothelioma: an overview and update on a rare vascular tumor. Oncol Rev. 2014 Oct 13;8(2):259. doi: 10.4081/oncol.2014.259. eCollection 2014 Sep 23. PMID 25992243
- [Background] Antonescu CR, Le Loarer F, Mosquera JM, Sboner A, Zhang L, Chen CL, Chen HW, Pathan N, Krausz T, Dickson BC, Weinreb I, Rubin MA, Hameed M, Fletcher CD. Novel YAP1-TFE3 fusion defines a distinct subset of epithelioid hemangioendothelioma. Genes Chromosomes Cancer. 2013 Aug;52(8):775-84. doi: 10.1002/gcc.22073. Epub 2013 Jun 5. PMID 23737213
- [Background] Errani C, Zhang L, Sung YS, Hajdu M, Singer S, Maki RG, Healey JH, Antonescu CR. A novel WWTR1-CAMTA1 gene fusion is a consistent abnormality in epithelioid hemangioendothelioma of different anatomic sites. Genes Chromosomes Cancer. 2011 Aug;50(8):644-53. doi: 10.1002/gcc.20886. Epub 2011 May 16. PMID 21584898
- [Background] Lamar JM, Motilal Nehru V, Weinberg G. Epithelioid Hemangioendothelioma as a Model of YAP/TAZ-Driven Cancer: Insights from a Rare Fusion Sarcoma. Cancers (Basel). 2018 Jul 10;10(7):229. doi: 10.3390/cancers10070229. PMID 29996478
- [Background] Rosenbaum E, Jadeja B, Xu B, Zhang L, Agaram NP, Travis W, Singer S, Tap WD, Antonescu CR. Prognostic stratification of clinical and molecular epithelioid hemangioendothelioma subsets. Mod Pathol. 2020 Apr;33(4):591-602. doi: 10.1038/s41379-019-0368-8. Epub 2019 Sep 19. PMID 31537895
- [Background] Kitaichi M, Nagai S, Nishimura K, Itoh H, Asamoto H, Izumi T, Dail DH. Pulmonary epithelioid haemangioendothelioma in 21 patients, including three with partial spontaneous regression. Eur Respir J. 1998 Jul;12(1):89-96. doi: 10.1183/09031936.98.12010089. PMID 9701420
- [Background] Yousaf N, Maruzzo M, Judson I, Al-Muderis O, Fisher C, Benson C. Systemic treatment options for epithelioid haemangioendothelioma: the Royal Marsden Hospital experience. Anticancer Res. 2015 Jan;35(1):473-80. PMID 25550590
- [Background] Shiba S, Imaoka H, Shioji K, Suzuki E, Horiguchi S, Terashima T, Kojima Y, Okuno T, Sukawa Y, Tsuji K, Umemoto K, Asagi A, Todaka A, Ueno M, Ikeda M, Morizane C, Furuse J. Clinical characteristics of Japanese patients with epithelioid hemangioendothelioma: a multicenter retrospective study. BMC Cancer. 2018 Oct 19;18(1):993. doi: 10.1186/s12885-018-4934-0. PMID 30340559
- [Background] Agulnik M, Yarber JL, Okuno SH, von Mehren M, Jovanovic BD, Brockstein BE, Evens AM, Benjamin RS. An open-label, multicenter, phase II study of bevacizumab for the treatment of angiosarcoma and epithelioid hemangioendotheliomas. Ann Oncol. 2013 Jan;24(1):257-63. doi: 10.1093/annonc/mds237. Epub 2012 Aug 21. PMID 22910841
- [Background] Zheng Z, Wang H, Jiang H, Chen E, Zhang J, Xie X. Apatinib for the treatment of pulmonary epithelioid hemangioendothelioma: A case report and literature review. Medicine (Baltimore). 2017 Nov;96(45):e8507. doi: 10.1097/MD.0000000000008507. PMID 29137048
- [Background] Semenisty V, Naroditsky I, Keidar Z, Bar-Sela G. Pazopanib for metastatic pulmonary epithelioid hemangioendothelioma-a suitable treatment option: case report and review of anti-angiogenic treatment options. BMC Cancer. 2015 May 13;15:402. doi: 10.1186/s12885-015-1395-6. PMID 25967676
- [Background] Chevreau C, Le Cesne A, Ray-Coquard I, Italiano A, Cioffi A, Isambert N, Robin YM, Fournier C, Clisant S, Chaigneau L, Bay JO, Bompas E, Gauthier E, Blay JY, Penel N. Sorafenib in patients with progressive epithelioid hemangioendothelioma: a phase 2 study by the French Sarcoma Group (GSF/GETO). Cancer. 2013 Jul 15;119(14):2639-44. doi: 10.1002/cncr.28109. Epub 2013 Apr 15. PMID 23589078
- [Background] Maher ER, Robinson KN, Scoble JE, Farrimond JG, Browne DR, Sweny P, Moorhead JF. Prognosis of critically-ill patients with acute renal failure: APACHE II score and other predictive factors. Q J Med. 1989 Sep;72(269):857-66. PMID 2616731
- [Background] Radzikowska E, Szczepulska-Wojcik E, Chabowski M, Oniszh K, Langfort R, Roszkowski K. Pulmonary epithelioid haemangioendothelioma--interferon 2-alpha treatment--case report. Pneumonol Alergol Pol. 2008;76(4):281-5. PMID 18785134
- [Background] Stacchiotti S, Provenzano S, Dagrada G, Negri T, Brich S, Basso U, Brunello A, Grosso F, Galli L, Palassini E, Libertini M, Colia V, Gronchi A, Dei Tos AP, Crippa F, Morosi C, Pilotti S, Casali PG. Sirolimus in Advanced Epithelioid Hemangioendothelioma: A Retrospective Case-Series Analysis from the Italian Rare Cancer Network Database. Ann Surg Oncol. 2016 Sep;23(9):2735-44. doi: 10.1245/s10434-016-5331-z. Epub 2016 Jun 22. PMID 27334221
- [Background] Kollar A, Jones RL, Stacchiotti S, Gelderblom H, Guida M, Grignani G, Steeghs N, Safwat A, Katz D, Duffaud F, Sleijfer S, van der Graaf WT, Touati N, Litiere S, Marreaud S, Gronchi A, Kasper B. Pazopanib in advanced vascular sarcomas: an EORTC Soft Tissue and Bone Sarcoma Group (STBSG) retrospective analysis. Acta Oncol. 2017 Jan;56(1):88-92. doi: 10.1080/0284186X.2016.1234068. Epub 2016 Nov 14. PMID 27838944
- [Background] McDonnell DP, Norris JD. Connections and regulation of the human estrogen receptor. Science. 2002 May 31;296(5573):1642-4. doi: 10.1126/science.1071884. PMID 12040178
- [Background] Revankar CM, Cimino DF, Sklar LA, Arterburn JB, Prossnitz ER. A transmembrane intracellular estrogen receptor mediates rapid cell signaling. Science. 2005 Mar 11;307(5715):1625-30. doi: 10.1126/science.1106943. Epub 2005 Feb 10. PMID 15705806
- [Background] Zhou X, Wang S, Wang Z, Feng X, Liu P, Lv XB, Li F, Yu FX, Sun Y, Yuan H, Zhu H, Xiong Y, Lei QY, Guan KL. Estrogen regulates Hippo signaling via GPER in breast cancer. J Clin Invest. 2015 May;125(5):2123-35. doi: 10.1172/JCI79573. Epub 2015 Apr 20. PMID 25893606
- [Background] De Marco P, Bartella V, Vivacqua A, Lappano R, Santolla MF, Morcavallo A, Pezzi V, Belfiore A, Maggiolini M. Insulin-like growth factor-I regulates GPER expression and function in cancer cells. Oncogene. 2013 Feb 7;32(6):678-88. doi: 10.1038/onc.2012.97. Epub 2012 Mar 19. PMID 22430216
- [Background] Zuco V, Pasquali S, Tortoreto M, Brich S, Percio S, Dagrada GP, Colombo C, Sanfilippo R, Lauricella C, Gounder M, El Bezawy R, Barisella M, Dei Tos AP, Casali PG, Gronchi A, Stacchiotti S, Zaffaroni N. Selinexor versus doxorubicin in dedifferentiated liposarcoma PDXs: evidence of greater activity and apoptotic response dependent on p53 nuclear accumulation and survivin down-regulation. J Exp Clin Cancer Res. 2021 Mar 1;40(1):83. doi: 10.1186/s13046-021-01886-x. PMID 33648535
- [Background] Stacchiotti S, Zuco V, Tortoreto M, Cominetti D, Frezza AM, Percio S, Indio V, Barisella M, Monti V, Brich S, Astolfi A, Colombo C, Pasquali S, Folini M, Gounder MM, Pantaleo MA, Collini P, Dei Tos AP, Casali PG, Gronchi A, Zaffaroni N. Comparative Assessment of Antitumor Effects and Autophagy Induction as a Resistance Mechanism by Cytotoxics and EZH2 Inhibition in INI1-Negative Epithelioid Sarcoma Patient-Derived Xenograft. Cancers (Basel). 2019 Jul 19;11(7):1015. doi: 10.3390/cancers11071015. PMID 31331120
- [Background] Stacchiotti S, Tortoreto M, Baldi GG, Grignani G, Toss A, Badalamenti G, Cominetti D, Morosi C, Dei Tos AP, Festinese F, Fumagalli E, Provenzano S, Gronchi A, Pennacchioli E, Negri T, Dagrada GP, Spagnuolo RD, Pilotti S, Casali PG, Zaffaroni N. Preclinical and clinical evidence of activity of pazopanib in solitary fibrous tumour. Eur J Cancer. 2014 Nov;50(17):3021-8. doi: 10.1016/j.ejca.2014.09.004. Epub 2014 Sep 27. PMID 25269954
- [Background] Stacchiotti S, Tortoreto M, Bozzi F, Tamborini E, Morosi C, Messina A, Libertini M, Palassini E, Cominetti D, Negri T, Gronchi A, Pilotti S, Zaffaroni N, Casali PG. Dacarbazine in solitary fibrous tumor: a case series analysis and preclinical evidence vis-a-vis temozolomide and antiangiogenics. Clin Cancer Res. 2013 Sep 15;19(18):5192-201. doi: 10.1158/1078-0432.CCR-13-0776. Epub 2013 Jul 25. PMID 23888069

DOCUMENTS (1):
  • Study Protocol (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT06680401/Prot_001.pdf